CLINICAL TRIAL: NCT00748124
Title: A Prospective Multicenter Randomized Clinical Study to Evaluate the PleuraSeal Sealant System as an Adjunct to Standard Closure Techniques for Control of Visceral Pleural Air Leaks Following Elective Pulmonary Resection Via Open Thoracotomy
Brief Title: PleuraSeal Pivotal Study (US)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis results were not supportive of primary endpoint
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUN-06-001
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Open Thoracotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PleuraSeal Sealant Device (Experimental)
  Interventions: Device: PleuraSeal Sealant System; Procedure: Standard Tissue Closure Techniques
- Control (Other)
  Interventions: Procedure: Standard Tissue Closure Techniques

INTERVENTIONS:
Device: PleuraSeal Sealant System — Lung Sealant Device + standard tissue closing techniques (sutures/staples)
  Arms: PleuraSeal Sealant Device
Procedure: Standard Tissue Closure Techniques — Standard tissue closure techniques (sutures/ staples) alone

SUMMARY:
To evaluate the safety and effectiveness of Confluent Surgical's PleuraSeal Sealant System in the treatment and control of intra and postoperative air leaks following pulmonary resection via an open thoracotomy. The performance of the PleuraSeal Sealant System as an adjunct to conventional closure techniques (i.e. surgical staples or sutures) will be compared to conventional surgical techniques alone.

ELIGIBILITY:
Inclusion Criteria:

* Elective pulmonary lobectomy, segmental and/or wedge resection in one or more lobes via an open thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects remaining air leak free from time of skin closure to hospital discharge. | 75 days

CONTACTS AND LOCATIONS:
Locations (1):
- Confluent Surgical, Bedford, Massachusetts, United States